CLINICAL TRIAL: NCT04790110
Title: The Progression of Tooth Wear and Possible Risk Factors: a 7 Year Follow up
Brief Title: 7 Year Follow up Analysis on the Speed of Progression of Tooth Wear Using 3D Subtraction
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Bevordering Tandheelkundige Kennis of the Nederlands Tijdschrift voor Tandheelkunde (Unknown)
Responsible Party: Sponsor
Other Study IDs: NTWP-ESOA2020
Record Dates: First submitted 2021-02-09; First posted 2021-03-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2022-10

CONDITIONS: Tooth Wear; Reflux Acid; Bruxism
Keywords: Progression of tooth wear
MeSH Terms: conditions — Tooth Wear; Gastroesophageal Reflux; Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Studie A ESO - monitoring: Patients that present themselves at the clinic through referral from their dentist with tooth wear, who have no request for help, receive a non-restorative 'counseling & monitoring' strategy , in which appropriate preventive measures are recommended and wear and tear is monitored and recorded by periodically taking intra-oral photographs and 3D scans

SUMMARY:
Prospective observational study with 7-year follow up. 55 patients are included with moderate to severe tooth wear, whereby through informed consent the decision was taking to monitor the patients. At the baseline and 1, 3 5, and the 7-year recall digital 3D scans will be made, which will be compared and subtracted.

DETAILED DESCRIPTION:
Prospective observational study with 7-year follow up. 55 patients are included with moderate to severe tooth wear, whereby through informed consent the decision was taking to monitor the patients. At the baseline and the 5-year recall digital 3D scans will be made, which will be compared and subtracted. Per tooth the loss of material is measured in maximum loss in height (µm) and volume (mm3) per year, using best fit alignment and 3D subtraction.

The loss of tooth material will be analyzed using descriptive statistics and possible effects of jaw type, tooth type and cusp type will be analyzed using multi level regression models.

The use of index teeth will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Generalized tooth wear
* A minimum of three posterior teeth (premolars and molars) per quadrant
* A maximum of one edentulous space in need for treatment, with a maximum span of one tooth-width

Exclusion Criteria:

* ASA 4
* Edentulous space has a span exceeding 1 tooth-width, or more than one space
* Functional problems (mouth opening <5cm, Temporomandibular Dysfunction)
* Severe periodontitis
* Strong gag reflex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants in this research will be drawn from the RTWP (Radboud Tooth Wear Project) patient sample which consists of nearly 200 tooth wear patients. Patients are included through dentist referral or of their own volition. Out of this population, 55 patients are managed non-restoratively, because they do not experience problems in regards to their tooth wear, and have no restorative treatment need in their perception
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2011-03-03 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
degree of dental wear in height | 7 years
  µm per year

SECONDARY OUTCOMES:
The use of index teeth | 7 years
  ICC correlation between ranking of patients according to whole dentition or index teeth

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed KE, Whitters J, Ju X, Pierce SG, MacLeod CN, Murray CA. Clinical Monitoring of Tooth Wear Progression in Patients over a Period of One Year Using CAD/CAM. Int J Prosthodont. 2017 Mar/Apr;30(2):153-155. doi: 10.11607/ijp.4990. PMID 28267825
- [Background] Loomans B, Opdam N, Attin T, Bartlett D, Edelhoff D, Frankenberger R, Benic G, Ramseyer S, Wetselaar P, Sterenborg B, Hickel R, Pallesen U, Mehta S, Banerji S, Lussi A, Wilson N. Severe Tooth Wear: European Consensus Statement on Management Guidelines. J Adhes Dent. 2017;19(2):111-119. doi: 10.3290/j.jad.a38102. PMID 28439579
- [Derived] Bronkhorst H, Bronkhorst E, Kalaykova S, Pereira-Cenci T, Huysmans MC, Loomans B. Inter- and intra-variability in tooth wear progression at surface-, tooth- and patient-level over a period of three years: A cohort study: Inter- and intra-variation in tooth wear progression. J Dent. 2023 Nov;138:104693. doi: 10.1016/j.jdent.2023.104693. Epub 2023 Sep 6. PMID 37683799